CLINICAL TRIAL: NCT06646133
Title: Machine Learning and 3D Image-Based Modeling for Real-Time Body Weight and Body Composition Estimation During Emergency Medical Care: Study 2 - Measure the Accuracy and Speed of Weight Estimations Using a 3D Camera System During Simulated Medical Emergencies
Brief Title: Machine Learning and 3D Image-Based Modeling for Real-Time Body Weight and Body Composition Estimation During Emergency Medical Care: Study 2
Status: Withdrawn | Type: Observational
Why Stopped: No funding received.
Sponsor: Florida Atlantic University (Other)
Responsible Party: Sponsor
Other Study IDs: 1791994(2)
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Body Weights and Measures; Body Weight in the Overweight and Obese Class - I Population; Weight Estimation; Emergency Drug Dosing
Keywords: weight estimation; emergency drug dosing; 3D camera; computer vision
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard care weight estimation: Simulated patients in whom standard methods of weight estimation will be used.
  Interventions: Diagnostic Test: Standard methods of weight estimation
- 3D camera weight estimation: Simulated patients in whom 3D camera estimates of weight will be used.
  Interventions: Diagnostic Test: 3D camera weight estimate

INTERVENTIONS:
Diagnostic Test: 3D camera weight estimate — Weight estimation using 3D camera system
  Groups: 3D camera weight estimation
Diagnostic Test: Standard methods of weight estimation — Standard methods of weight estimation will be used
  Groups: Standard care weight estimation

SUMMARY:
The goal of this prospective crossover simulation study is to evaluate the accuracy and usability of a 3D camera weight estimation system during simulated emergency care in adult simulated patients, when used by emergency physicians. The main questions the study aims to answer are:

* to evaluate the accuracy of 3D camera weight estimation during simulated emergency care, when compared with standard methods
* to evaluate the usability of 3D camera weight estimation during emergency care, when compared with standard methods
* to evaluate the inter-user reliability of 3D camera weight estimates Volunteers for simulated patients will be required to have anthropometric measurements, a DXA scan, and 3D camera weight estimates.

Physician volunteers will need to participate in simulated emergency scenarios during which weight-based therapy must be administered.

There will be no interventions.

DETAILED DESCRIPTION:
The performance of the 3D camera system needs to be evaluated in conditions in which it will be used in a clinical setting, but without the risk to patients. It also needs to be compared against other, standard, methods of weight estimation. In addition the downstream accuracy of drug doses, with the correct use of alternative dose scalars (such as ideal body weight or lean body weight) in patients with obesity needs to be evaluated.

In this prospective crossover simulation study, resident and attending emergency physician volunteers will conduct simulated emergency care on simulated patient volunteers. The physicians will be randomised to start with either 3D camera systems, or standard care systems. After completing the scenario they will perform a new simulation scenario on a different patient using standard methods of weight estimation (crossover). At the end of the data collection session, each physician will have performed four scenarios (two standard methods, two 3D camera methods). Each simulated patient will similarly have participated in two standard method scenarios and two 3D camera scenarios. Each simulated patient and each physician will only have a single encounter.

In this way the accuracy of weight estimation and drug dosing can be compared between the 3D camera system and standard methods. In addition, inter-rater reliability can be determined and compared between resident and attending physicians.

ELIGIBILITY:
Inclusion Criteria for simulated patients:

* Any volunteer aged ≥18 years.

Exclusion Criteria for simulated patients:

* Participants with a body weight exceeding the DXA machine capacity >204kg (450lbs);
* Pregnant participants; participants with medical conditions that could confound the study;
* Participants with any metallic surgical implants;
* Participants who have had an x-ray with contrast in the past week;
* Participants who have taken calcium supplements in the 24 hours prior to the study.

Inclusion criteria for Emergency Physicians:

- Any willing emergency medicine resident or attending physician.

Exclusion criteria for Emergency Physicians:

- Any physical limitation to performing anthropometric measurements as part of simulation scenario.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Simulated patients will be enrolled from students, staff and faculty at the Boca Raton campus of Florida Atlantic university.
  Emergency physician participants will be enrolled from resident and attending emergency physicians in south Florida.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2027-07-01 (Estimated); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Weight estimation accuracy | During the simulation (intervention) procedure
  The accuracy of estimations of total body weight, ideal body weight and lean body weight will be compared against ground truth data, and against other weight estimation systems.
Weight estimation time | During the simulation (intervention) procedure
  The time taken to obtain a weight estimate will be compared against other weight estimation systems.
Drug dose accuracy | During the simulation (intervention) procedure
  The accuracy of drug doses calculated using estimated weight will be compared against a ground truth value, and compared with other weight estimation systems.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida Atlantic University, Boca Raton, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
The data will be made available on request.
Supporting Information: Study Protocol
Time Frame: Within 6 months after the completion of the study.

REFERENCES:
- [Background] Wells M, Goldstein L. Appropriate Statistical Analysis and Data Reporting for Weight Estimation Studies. Pediatr Emerg Care. 2023 Jan 1;39(1):62-63. doi: 10.1097/PEC.0000000000002862. Epub 2022 Oct 1. No abstract available. PMID 36190388
- [Background] Wells M, Goldstein LN, Cattermole G. Development and Validation of a Length- and Habitus-Based Method of Ideal and Lean Body Weight Estimation for Adults Requiring Urgent Weight-Based Medical Intervention. Eur J Drug Metab Pharmacokinet. 2022 Nov;47(6):841-853. doi: 10.1007/s13318-022-00796-3. Epub 2022 Sep 19. PMID 36123560
- [Background] Wells M, Goldstein LN. Estimating Lean Body Weight in Adults With the PAWPER XL-MAC Tape Using Actual Measured Weight as an Input Variable. Cureus. 2022 Sep 17;14(9):e29278. doi: 10.7759/cureus.29278. eCollection 2022 Sep. PMID 36277563
- [Background] Wells M, Henry B, Goldstein L. Weight Estimation for Drug Dose Calculations in the Prehospital Setting - A Systematic Review. Prehosp Disaster Med. 2023 Aug;38(4):471-484. doi: 10.1017/S1049023X23006027. Epub 2023 Jul 13. PMID 37439214
- [Background] Wells M, Goldstein LN, Alter SM, Solano JJ, Engstrom G, Shih RD. The accuracy of total body weight estimation in adults - A systematic review and meta-analysis. Am J Emerg Med. 2024 Feb;76:123-135. doi: 10.1016/j.ajem.2023.11.037. Epub 2023 Nov 29. PMID 38056057
- [Background] Wells M, Goldstein LN, Wells T, Ghazi N, Pandya A, Furht B, Engstrom G, Jan MT, Shih R. Total body weight estimation by 3D camera systems: Potential high-tech solutions for emergency medicine applications? A scoping review. J Am Coll Emerg Physicians Open. 2024 Oct 4;5(5):e13320. doi: 10.1002/emp2.13320. eCollection 2024 Oct. PMID 39371964